CLINICAL TRIAL: NCT04866589
Title: The Effectiveness of Distributing Free Face Masks to Increase Use of Face Masks During the COVID-19 Pandemic. A Randomised Experiment in Stovner District, Oslo, Norway
Brief Title: COVID-19: The Effectiveness of Free Face Mask Distribution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: Stovner District, City of Oslo, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: FaceMaskRCT Stovner
Record Dates: First submitted 2021-04-15; First posted 2021-04-30 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Face masks; Infection control; Behavioral intervention
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: The team members from the Stovner district-administration will send a numbered list to Norwegian Institute of Public Health-team, with the names of the stores. The ordering of the stores will define the numbers used to represent each store in the randomisation process. Using Stata software, we will carry out 13 separate and independent randomisations, each assigning the intervention to half the included stores. An additional randomisation to the treatment or control group will be carried out for a marginal store each day in the event of an odd number of stores.
  Unless it proves too logistically cumbersome, we will also randomise the corona hosts, i.e. the store they are allocated to will be decided through randomisation.
Masking Description: The analyst will receive a dataset in a format which makes it impossible for him/her to know which of the two arms in the dataset represents intervention or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distribution of free face masks (Experimental): Face masks will be handed out for free to all customers entering the grocery stores.
  Interventions: Behavioral: Distribution of free face masks
- Control (No Intervention): Business as usual.

INTERVENTIONS:
Behavioral: Distribution of free face masks — "Corona hosts" will be placed at the entrance of the intervention stores, and hand out face masks to customers entering the store.
  Arms: Distribution of free face masks

SUMMARY:
The investigators will carry out a randomised trial of free face mask distribution in Stovner District, Oslo, Norway. Ten grocery stores will serve as study sites. Over three weeks the stores will be randomised daily to having "corona hosts" outside their entrance, handing out face masks to customers. The investigators will compare the proportion of customers who wear face masks as they enter the store in stores with or without face mask distribution.

ELIGIBILITY:
All grocery stores in the Stovner district are eligible as long as they have not, or only sporadically, had free distribution of face masks previously.

At the customer level, we will only include those 12 years or older (age based on the outcome assessor's judgement).

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Face mask use | Through study completion, 3 weeks.
  Proportion of customers wearing a face mask

SECONDARY OUTCOMES:
Correct use of face masks | Through study completion, 3 weeks
  Proportion of customers wearing a face mask correctly (i.e. covering mouth and nose)

CONTACTS AND LOCATIONS:
Overall Officials: Atle Fretheim, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Stover District, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the full dataset as soon as it as ready. All data are anonymous, so there are no person data issues to take into consideration.
Supporting Information: Study Protocol, Analytic Code
Time Frame: From early June 2021, and for all foreseeable future.
Access Criteria: None - anyone will have access to the dataset.

REFERENCES:
- [Derived] Elgersma IH, Fretheim A, Indseth T, Munch AT, Johannessen LB, Hansen CE. The Evaluation of a Social Media Campaign to Increase COVID-19 Testing in Migrant Groups: Cluster Randomized Trial. J Med Internet Res. 2022 Mar 24;24(3):e34544. doi: 10.2196/34544. PMID 35285811